CLINICAL TRIAL: NCT01522118
Title: Focal Therapy With Magnetic Resonance Guided Focused Ultrasound Treatment of Locally Non-Advanced Prostate Cancer: Phase 1 Study
Brief Title: MR-guided Focused Ultrasound Treatment of Prostate Cancer: Focal Therapy for Locally Non-Advanced Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Alessandro Napoli, Assistant Professor, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PCa-MRgFUS-I
Record Dates: First submitted 2012-01-23; First posted 2012-01-31 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; High Intensity Focused Ultrasound; Magnetic Resonance guided Focused Ultrasound; Non-invasive therapy; Focal Disease
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIFU (Experimental): (high intensity focused ultrasound)
  Interventions: Device: ExAblate 2100; InSightec

INTERVENTIONS:
Device: ExAblate 2100; InSightec — Patients with biopsy proven locally non-advanced T2 prostate cancer identified at 3T MR examination including dynamic contrast enhanced (DCE-with time to peak and mean transit time evaluation) and candidate to radical prostatectomy will undergo Magnetic Resonance guided Focused Ultrasound (MRgFUS) ablation. The procedure is carried out either under general anesthesia or spinal block.
  MR images allow correct identification of the target as well as vital structure to avoid during energy delivery. Treatment safety and efficacy is monitored in real time using MR thermometry. Adjustments of energy direction and intensity can be made according to the real time monitoring. Pre- and post-ablative MR examinations will serve to analyze differences of DCE features of the neoplastic tissue; therapy-induced alterations will also be compared to histopathology findings from whole section prostate specimens

SUMMARY:
Since prostate specific antigen (PSA) was introduced as a clinical screening tool for prostate cancer, more men are diagnosed with small foci of cancers instead of the advanced disease. The present choice of treatment for men with localized prostate cancer lies between active surveillance and radical therapy. Thus, the option of treating only the cancer within the prostate gland and sparing the non-cancerous tissue is quite appealing, yet very controversial. At present there are no consistent scientific data on focal therapy and its major effectiveness.

Focal therapy for prostate cancer is defined as therapy that selectively ablates known disease while preserving existing functions, with the overall aim of minimizing lifetime morbidity without compromising life expectancy.

The aim of the investigators study is to test if Magnetic Resonance guided Focused Ultrasound ablation can determine non-invasive necrosis of focal, locally non-advanced prostate cancer.

The study i designed as Phase 1, treatment & resection protocol. With this project the investigators further aim to evaluate the safety and identify side effects of Magnetic Resonance guided Focused Ultrasound in treating focal prostate cancer.

This design will also expand knowledge of the effect of Magnetic Resonance guided Focused Ultrasound onto peri-prostatic environment and to determine if surgery can safely be adopted after this non-invasive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient of age between 40 to 85
* Patient with organ-confined Pca (cT1c and cT2a, N0, M0), diagnosed with TRUS biopsy (min:12 cores)
* Patient with PSA ≤ 10 ng/mL
* Gleason score 6 (3+3) or max 7 (3+4)
* Up to two (2) MR identifiable lesions
* No definite evidence of extracapsular extension

Exclusion Criteria:

* Patient under medications that can affect PSA for the last 3 months prior to MRgFUS treatment (Androgen Deprivation Treatment; alpha reductase inhibitors)
* Any rectal pathology, anomaly or previous treatment
* Identified calcification of 2 mm or more in largest diameter neighboring the rectal wall
* Bladder cancer
* Seminal vesicle/lymph node
* Prostate with multiple cystic lesions

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety | One year
  Measure of expected or UN-expected adverse events

SECONDARY OUTCOMES:
Efficacy | 18 months
  Measure of ablated area in terms of necrosis vs residual tumor

CONTACTS AND LOCATIONS:
Overall Officials: alessandro napoli, MD, PhD, Principal Investigator — Department of Radiological Sciences, Sapienza University of Rome
Locations (1):
- Department of Radiological Sciences, Sapienza University of Rome, Rome, Italy